CLINICAL TRIAL: NCT02650297
Title: The Effect of Combined Decongestive Therapy and Pneumatic Compression Pump on Body Image in Patients With Lymphedema Secondary to Breast Cancer Treatment
Brief Title: The Effect of Combined Decongestive Therapy and Pneumatic Compression Pump on Body Image in Patients With Lymphedema
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: badri jaafari (Other)
Responsible Party: Sponsor-Investigator, badri jaafari, faculty member of IAUKazeroun, Islamic Azad University, Kazeroun
Organization: Islamic Azad University, Kazeroun (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IAUKazeroun
Record Dates: First submitted 2015-12-29; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Lymphedema
Keywords: Lymphedema secondary to breast cancer; Breast cancer; Body image
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDT and pneumatic compression pump (Experimental): combined decongestive therapy consists of the pressure of bandage, manual lymphatic drainage, and exercises that increase the flow of lymph and skin care are used. Intermittent pneumatic pump is not as a part of CDT, but it can be used as an adjunct method. This device according to a specific program is air filled and emptied. The device leads the lymphatic fluid from distal to the proximal part of extremities and then to the trunk.
  Interventions: Other: combined decongestive therapy; Device: pneumatic compression pump
- not CDT and pneumatic compression pump (No Intervention): Patients in the control group received no treatment for lymphedema but were placed on the waiting list for CDT as soon as possible after the 8 weeks follow-up period.

INTERVENTIONS:
Other: combined decongestive therapy — Patients in the intervention group received treatment with combined decongestive therapy and pneumatic compression pump. Patients in the control group received no treatment for lymphedema but were placed on the waiting list for combined decongestive therapy and pneumatic compression pump as soon as possible after the 8 weeks follow-up period.
  Arms: CDT and pneumatic compression pump
Device: pneumatic compression pump — Intermittent pneumatic pump or pressure therapy is not as a part of CDT, but it can be used as an adjunct method. This device intermittently and according to a specific program is air filled and emptied. The device leads the lymphatic fluid from distal to the proximal part of extremities and then to the trunk
  Arms: CDT and pneumatic compression pump

SUMMARY:
Patients with lymphedema may experience pain and body image issues. This study investigates the effect of Combined Decongestive Therapy and pneumatic compression pump on body image in patients with lymphedema secondary to breast cancer treatment.42 women with breast cancer related lymphedema participated. All patients completed the body image and relationships scale. Researchers divided the participants randomly into an intervention (n=21) or control group (n=21). In the first phase, CDT was accompanied by use of a compression pump for four weeks, three days per week. In the second phase, Combined DecongestiveTherapy was performed daily without compression pump for four weeks by patients at home. At the end of each phase, both groups completed the questionaire. Researchers analyzed the data with SPSS v.17.

DETAILED DESCRIPTION:
Background:

Lymphedema is a common complication for breast cancer therapy. Patients with lymphedema may experience pain and body image issues. This study investigates the effect of Combined Decongestive Therapy and pneumatic compression pump on body image in patients with lymphedema secondary to breast cancer treatment.

methods: 42 women with breast cancer related lymphedema participated. All patients completed the body image and relationships scale. Researchers divided the participants randomly into an intervention (n=21) or control group (n=21). A certified nurse worked on Combined Decongestive Therapy in the intervention group in two phases. In the first phase, CDT was accompanied by use of a compression pump for four weeks, three days per week. In the second phase, CDT was performed daily without compression pump for four weeks by patients at home. At the end of each phase, both groups completed the questionaire. Researchers analyzed the data with SPSS v.17.

ELIGIBILITY:
Inclusion criteria:

1. histoty of breast cancer,
2. history of surgery and chemotherapy and as needed hormone therapy and radiotherapy,
3. affected by lymphedema (with degree of mild to severe) based on specialist diagnosis,
4. at least 1 year ago was undergone axillary node dissection,
5. do not have knowledge about combined decongestive therapy,
6. phone accessibility,
7. 35-70 years old.

Exclusion criteria:

1. psychotic disorder,
2. existence sever pain at axillary area,
3. history of hysterectomy duo to uterus cancer,
4. severe cardiac disease,
5. heart failure,
6. renal failure,
7. severe hypertension,
8. existing other malignancies,
9. recurrent infection in arm,
10. musclo skeletal disease

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
changes in the body image | change from baseline body image at 8 weeks
  Body image evaluated with the body image and relationships scale. Body image and relationships scale is a questionnaire that consists of 32 items in the three subscales or factors, named strength and health, social barriers, and appearance and sexuality. Higher scores on each subscale indicated greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: badri jaafari, author, Study Chair — Department of Nursing, College of Nursing & Midwifery, Kazeroun Azad University, Kazeroun, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Isaksson G, Feuk B. Morbidity from axillary treatment in breast cancer--a follow-up study in a district hospital. Acta Oncol. 2000;39(3):335-6. doi: 10.1080/028418600750013104. No abstract available. PMID 10987230
- [Result] Kaviani A, Lotfi M. Control of lymphedema after breast cancer treatment. 1st ed. Tehran: Tehran university of medical
- [Result] Didem K, Ufuk YS, Serdar S, Zumre A. The comparison of two different physiotherapy methods in treatment of lymphedema after breast surgery. Breast Cancer Res Treat. 2005 Sep;93(1):49-54. doi: 10.1007/s10549-005-3781-2. PMID 16184458
- [Result] Nielsen I, Gordon S, Selby A. Breast cancer-related lymphoedema risk reduction advice: a challenge for health professionals. Cancer Treat Rev. 2008 Nov;34(7):621-8. doi: 10.1016/j.ctrv.2007.11.002. Epub 2008 Aug 8. PMID 18691823
- [Result] Hormes JM, Lytle LA, Gross CR, Ahmed RL, Troxel AB, Schmitz KH. The body image and relationships scale: development and validation of a measure of body image in female breast cancer survivors. J Clin Oncol. 2008 Mar 10;26(8):1269-74. doi: 10.1200/JCO.2007.14.2661. PMID 18323550
- [Result] Ridner SH. The psycho-social impact of lymphedema. Lymphat Res Biol. 2009;7(2):109-12. doi: 10.1089/lrb.2009.0004. PMID 19534633
- [Result] Pain SJ, Purushotham AD. Lymphoedema following surgery for breast cancer. Br J Surg. 2000 Sep;87(9):1128-41. doi: 10.1046/j.1365-2168.2000.01569.x. PMID 10971418
- [Result] Foldi M. Lymphology in the second millennium. Lymphology. 2001 Mar;34(1):12-21. No abstract available. PMID 11307660
- [Result] Harris SR, Hugi MR, Olivotto IA, Levine M; Steering Committee for Clinical Practice Guidelines for the Care and Treatment of Breast Cancer. Clinical practice guidelines for the care and treatment of breast cancer: 11. Lymphedema. CMAJ. 2001 Jan 23;164(2):191-9. PMID 11332311
- [Result] Uzkeser H, Karatay S, Erdemci B, Koc M, Senel K. Efficacy of manual lymphatic drainage and intermittent pneumatic compression pump use in the treatment of lymphedema after mastectomy: a randomized controlled trial. Breast Cancer. 2015 May;22(3):300-7. doi: 10.1007/s12282-013-0481-3. Epub 2013 Aug 8. PMID 23925581
- [Result] Irdesel J, Celiktas SK. Effectiveness of exercise and compression garments in the treatment of breast cancer related lymphedema- Original article. Turk J Phys Med Rehab, 2007;53:16-21.
- [Result] Passik S, Newman M, Brennan M, Holland J. Psychiatric consultation for women undergoing rehabilitation for upper-extremity lymphedema following breast cancer treatment. J Pain Symptom Manage. 1993 May;8(4):226-33. doi: 10.1016/0885-3924(93)90132-f. PMID 7963764
- [Result] Pruzinsky T. Enhancing quality of life in medical populations: a vision for body image assessment and rehabilitation as standards of care. Body Image. 2004 Jan;1(1):71-81. doi: 10.1016/S1740-1445(03)00010-X. PMID 18089142
- [Result] Passik SD, McDonald MV. Psychosocial aspects of upper extremity lymphedema in women treated for breast carcinoma. Cancer. 1998 Dec 15;83(12 Suppl American):2817-20. doi: 10.1002/(sici)1097-0142(19981215)83:12b+3.0.co;2-2. PMID 9874404
- [Result] Speck RM, Gross CR, Hormes JM, Ahmed RL, Lytle LA, Hwang WT, Schmitz KH. Changes in the Body Image and Relationship Scale following a one-year strength training trial for breast cancer survivors with or at risk for lymphedema. Breast Cancer Res Treat. 2010 Jun;121(2):421-30. doi: 10.1007/s10549-009-0550-7. Epub 2009 Sep 22. PMID 19771507
- [Result] Poorkiani M, Abbaszadeh A, Hazrati M, Jafari P, Sadeghi M, Mohammadianpanah M. The effect of rehabilitation on quality of life in female breast cancer survivors in Iran. Indian J Med Paediatr Oncol. 2010 Oct;31(4):105-9. doi: 10.4103/0971-5851.76190. PMID 21584214
- [Result] Teo I, Novy DM, Chang DW, Cox MG, Fingeret MC. Examining pain, body image, and depressive symptoms in patients with lymphedema secondary to breast cancer. Psychooncology. 2015 Nov;24(11):1377-83. doi: 10.1002/pon.3745. Epub 2015 Jan 20. PMID 25601235
- See also: website — http://www.tums.ac.ir/faculties/akaviani
- See also: Text Link — http://www.ncbi.nlm.nih.gov/pubmed/16184458
- See also: Text Link — http://www.ncbi.nlm.nih.gov/pubmed/18691823
- See also: Text Link — http://www.ncbi.nlm.nih.gov/pubmed/18323550
- See also: Text Link — http://www.ncbi.nlm.nih.gov/pubmed/11307660
- See also: Text Link — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC80678/
- See also: Text Link — http://www.ncbi.nlm.nih.gov/pubmed/23925581
- See also: Text Link — http://www.ncbi.nlm.nih.gov/pubmed/7963764
- See also: Text Link — http://www.ncbi.nlm.nih.gov/pubmed/18089142
- See also: Text Link — http://www.ncbi.nlm.nih.gov/pubmed/9874404
- See also: Text Link — http://www.ncbi.nlm.nih.gov/pubmed/19771507
- See also: Text Link — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3089917/